CLINICAL TRIAL: NCT02477046
Title: Assessment of Community Transmission of Sabin Type 2 Virus in Bangladesh
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Virginia (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Mami Taniuchi, PhD, Assistant Professor of Research, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00000447; PR-15004 (Other: ICDDRB)
Record Dates: First submitted 2015-06-18; First posted 2015-06-22 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Vaccine Virus Shedding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- tOPV + IPV (Experimental): tOPV (6, 10, and 14 weeks) + IPV (14 weeks) Randomized to receive tOPV plus IPV boost
  Interventions: Biological: tOPV; Biological: IPV
- bOPV + IPV (Experimental): bOPV (6, 10, and 14 weeks) + IPV (14 weeks) Randomized to receive bOPV plus 1 IPV boost
  Interventions: Biological: bOPV; Biological: IPV
- bOPV + 2 IPV (Experimental): bOPV (6, 10, and 14 weeks) + IPV (14 and 18 weeks) Randomized to receive bOPV plus 2 IPV boost
  Interventions: Biological: bOPV; Biological: IPV

INTERVENTIONS:
Biological: tOPV — administered per protocol
  Arms: tOPV + IPV
Biological: bOPV — administered per protocol
  Arms: bOPV + 2 IPV; bOPV + IPV
Biological: IPV — administered per protocol

SUMMARY:
The Strategic Advisory Group of Experts on Immunization (SAGE) has set a plan to replace trivalent oral polio vaccine (tOPV) with bivalent OPV (bOPV) plus inactivated polio vaccine (IPV) in routine immunization globally, to be instituted in 2015-2016. At the community level, the impact of the change from tOPV + IPV to bOPV + IPV on Sabin virus fecal-oral transmission (duration of circulation, degree of genetic reversion) and the persistence of environmental contamination are unknown. Also unknown is the impact of the change from tOPV to bOPV on community circulation of Sabin 2 after a special immunization (SI) activity with monovalent oral poliovirus type 2 (mOPV2). Finally it is unknown at the level of an individual child if type 2 fecal shedding will be limited by cross-protection from oral vaccination with Sabin type 1 and 3.

The investigators propose to measure at a community level transmission of Sabin 2 virus in Bangladesh, a low income country, where fecal-oral transmission and environmental exposures are high, comparing transmission in the setting of vaccination with tOPV+IPV vs. bOPV+IPV. The study will be conducted in 67 villages in Matlab, Bangladesh, using a cluster-randomized study design. Villages in Matlab will be randomly assigned to receive as part of routine immunization (RI) activities: (1) tOPV (6,10,14 weeks) plus IPV at 14 weeks; (2) bOPV (6,10, 14 weeks) plus IPV at 14 weeks; or (3) bOPV (6,10, 14 weeks) plus IPV at 14 and 18 weeks. Community and environmental surveillance for Sabin 2 virus will be conducted in each village over the 9 month period of these RI activities. In addition, a SI activity with mOPV2 will occur 9 months into the study to model an outbreak response. For the 6 months following the mOPV2 challenge, the impact of the different vaccination regimens on Sabin 2 transmission in the community will be determined, as well as individual level protection (as measured by fecal shedding from days 7-70 after mOPV2 challenge).

ELIGIBILITY:
Inclusion Criteria:

* A male or female infant at least 6 weeks of age (42-48 days) at the time of enrollment
* For the Special Immunization Activity (SIA) only, being age 5 years or younger at the time of the SIA
* An infant whose parent or guardian's primary residence, at the time of first Expanded Program on Immunization (EPI) vaccinations, is a village selected to receive polio vaccine.
* Written informed consent obtained from the parent or guardian of the participant, prior to the participants's first study vaccination

Exclusion Criteria:

* History of prior polio vaccination (in the 810 infants enrolled at 6 weeks of age only)
* Hypersensitivity to the active substance or any component in the vaccine
* Subjects with uncorrected congenital malformation
* Infants with known or suspected immunodeficiency

Ages: 42 Days to 48 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 810 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-07 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
fecal shedding of type 2 Sabin virus by quantitative reverse transcription polymerase chain reaction (RT-qPCR) in 60% of infants that did not receive the mOPV2 challenge | 10 weeks following mOPV2 challenge at month 9 of the study
  The transmission rate of type 2 Sabin virus in the 60% of the enrolled infants that did not receive the mOPV2 challenge between Arm A vs Arm B, Arm A vs Arm C, and Arm B and Arm C.

SECONDARY OUTCOMES:
fecal shedding of type 2 Sabin virus by RT-qPCR in 40% of infants that received the mOPV2 challenge | 10 weeks following mOPV2 challenge at month 9 of the study
  Individual protection to type 2 poliovirus from different vaccination schedules

CONTACTS AND LOCATIONS:
Overall Officials: William A Petri, Jr., MD, PhD, Principal Investigator — University of Virginia; Mami Taniuchi, PhD, Principal Investigator — University of Virginia; K Zaman, MBBS, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Matlab, Bangladesh

REFERENCES:
- [Background] Taniuchi M, Begum S, Uddin MJ, Platts-Mills JA, Liu J, Kirkpatrick BD, Chowdhury AH, Jamil KM, Haque R, Petri WA Jr, Houpt ER. Kinetics of poliovirus shedding following oral vaccination as measured by quantitative reverse transcription-PCR versus culture. J Clin Microbiol. 2015 Jan;53(1):206-11. doi: 10.1128/JCM.02406-14. Epub 2014 Nov 5. PMID 25378579
- [Derived] Famulare M, Wong W, Haque R, Platts-Mills JA, Saha P, Aziz AB, Ahmed T, Islam MO, Uddin MJ, Bandyopadhyay AS, Yunus M, Zaman K, Taniuchi M. Multiscale model for forecasting Sabin 2 vaccine virus household and community transmission. PLoS Comput Biol. 2021 Dec 21;17(12):e1009690. doi: 10.1371/journal.pcbi.1009690. eCollection 2021 Dec. PMID 34932560
- [Derived] Taniuchi M, Famulare M, Zaman K, Uddin MJ, Upfill-Brown AM, Ahmed T, Saha P, Haque R, Bandyopadhyay AS, Modlin JF, Platts-Mills JA, Houpt ER, Yunus M, Petri WA Jr. Community transmission of type 2 poliovirus after cessation of trivalent oral polio vaccine in Bangladesh: an open-label cluster-randomised trial and modelling study. Lancet Infect Dis. 2017 Oct;17(10):1069-1079. doi: 10.1016/S1473-3099(17)30358-4. Epub 2017 Jul 7. PMID 28693854
- Available data/document: Statistical Analysis Plan — https://idmod.sharepoint.com/projects/_layouts/15/guestaccess.aspx?guestaccesstoken=3%2bxJO%2bcBwXx6PfMuzCQmu8ESB0X7mhLPtowTTLaYTmY%3d&docid=02ab39752ccb14c10bdfd61c0a731e6ff&rev=1